CLINICAL TRIAL: NCT05586321
Title: A First-in-Human, Open-label, Dose-finding Trial to Evaluate the Safety and Antitumor Activity of GEN1056 in Subjects With Advanced Solid Tumors
Brief Title: Study of Safety and Antitumor Activity of GEN1056 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1056-01; 2022-001003-40 (EudraCT Number); 2024-514357-29-00 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2022-10-11; First posted 2022-10-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor, Adult
Keywords: Cancer; Advanced cancer; Phase I; Metastatic cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GEN1056 Monotherapy (Experimental)
  Interventions: Biological: GEN1056

INTERVENTIONS:
Biological: GEN1056 — GEN1056 will be administered as an intravenous (IV) infusion. The dose levels will be determined by the starting dose and the escalation steps taken in the trial in Part 1. In Part 2, the dose and schedule will be decided based on data outcome from Part 1.

SUMMARY:
The main purpose of this first-in-human study of GEN1056, is to evaluate safety. In addition, the study will determine the recommended dose and frequency for subsequent clinical studies and will assess the preliminary anti-tumor activity of GEN1056. GEN1056 will be studied in patients with advanced or metastatic solid cancer, for whom standard of care (SOC) therapy is not an option. All participants will get GEN1056.

DETAILED DESCRIPTION:
The trial is a first-in-human open-label, dose-finding, multinational safety trial, in participants with advanced or metastatic solid (non central nervous system [CNS]) tumors that have exhausted SOC therapy or are not candidates for SOC therapy, evaluating the safety, tolerability, preliminary antitumor activity, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of GEN1056.

The trial will be conducted as follows:

* The Dose Escalation part (Part 1) will explore the safety of escalating doses of GEN1056
* The Dose schedule optimization part (Part 2) will explore further safety and tolerability in an alternate schedule of a dose based on data outcome available from Part 1.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with histologically or cytologically confirmed non-CNS advanced or metastatic solid tumors which has progressed despite standard therapy, or subjects who are intolerant of standard therapy, or for which no standard therapy exists, and for whom, in the opinion of the investigator, experimental therapy with GEN1056 may be beneficial
* Have personally (or in countries where permitted, their legally acceptable representative) signed an Informed Consent Form (ICF)
* Are at least 18 years of age.
* Have measurable disease according to the RECIST v1.1 criteria.
* Have an ECOG PS of 0 to 1 at screening and on C1D1 pre-treatment.
* Have acceptable laboratory test results during the screening period.
* Must provide an archival (FFPE) tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated.
* A female subject with reproductive potential must agree to use adequate contraception during the trial, and for 4 months after receiving the last dose of trial drug GEN1056.

Key Exclusion Criteria:

* Subject is considered a poor medical risk due to a serious, uncontrolled inter-current illness
* Prior therapy with a checkpoint inhibitor agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor.
* Prior exposure to any of the following prior therapies within the specified timeframes:

  1. Systemic cytotoxic chemotherapy or antineoplastic biological therapy within 28 days or at least 5 elimination half-lives of the drug (whichever is shorter) of the first dose of trial treatment
  2. Radiotherapy within 21 days of start of trial treatment. Note: palliative radiotherapy be allowed.
  3. Prior treatment with live, attenuated vaccines within 28 days prior to initiation of GEN1056
* Known active CNS metastases and/or carcinomatous meningitis, or spinal cord compression.
* Positive for Human Immunodeficiency Virus (HIV), Hepatitis B (Hepatitis B Surface Antigen (HBsAg), HBV DNA), or Hepatitis C infection (Hepatitis C Virus Ribonucleic Acid (HCV RNA), HCV antibodies).
* An active, known, or suspected autoimmune disease, requiring systemic steroid.
* A condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first treatment.
* History of non-infectious pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease requiring treatment with steroids.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | DLTs are evaluated during the first 21 days after a patient's first dose
  To define the maximum tolerated dose (MTD) and/or recommended phase 2 dose(s) (RP2D) of GEN1056
Incidence and severity of adverse events (AEs) | Throughout the trial until the end of the safety follow-up period (90 days after last dose)
Number of participants with clinical significant shifts from baseline in clinical laboratory parameters | Throughout the trial until the end of the safety follow-up period (90 days after last dose)
  Clinical laboratory parameters assessed: Hematology, biochemistry, coagulation, TSH, T3 and T4, urinalysis

SECONDARY OUTCOMES:
Objective response rate (ORR) | From first infusion of trial drug to the last evaluable imaging assessment (an estimated average of 7 months)
  Anti-tumor activity of GEN1056 as monotherapy according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for responders (with confirmation)
Duration of response (DOR) | From initial onset of response to first progression event (defined as radiographic progression or death; an estimated average of 7 months)
  Anti-tumor activity of GEN1056 as monotherapy according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for responders (with confirmation)
Progression-free survival (PFS) | From first infusion of trial drug to first progression event (defined as radiographic progression or death; an estimated average of 7 months)
  Anti-tumor activity of GEN1056 as monotherapy according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Overall survival (OS) | From first infusion of trial drug to death due to any cause, or to last contact date in case of no observed death (assessed up to 2 years after the last participant's first dose in the trial)
  Defined as time of death, due to any cause
Rate at which the drug is removed from the body (clearance) | Throughout the trial until the end of the safety follow-up period (90 days after last dose)
Amount of drug in the body (volume of distribution) | Throughout the trial until the end of the safety follow-up period (90 days after last dose)
Area under the concentration time curve (AUC) from time zero to last quantifiable sample AUClast | Throughout the trial until the end of the safety follow-up period (90 days after last dose)
Maximum (peak) observed serum drug concentration (Cmax) | Throughout the trial until the end of the safety follow-up period (90 days after last dose)
Time to reach maximum (peak) serum drug concentration (Tmax) after dosing | Throughout the trial until the end of the safety follow-up period (90 days after last dose)
Time after dosing at which the lowest drug concentration is observed before the next dose is administered, predose trough concentration (Ctrough) | Throughout the trial until the end of the safety follow-up period (90 days after last dose)
Elimination half-life (T1/2) of the drug | Throughout the trial until the end of the safety follow-up period (90 days after last dose)
Incidence of anti-drug antibodies (anti GEN1056 antibodies) | Throughout the trial until the end of the safety follow-up period (90 days after last dose)
  Characterize the immunogenicity of GEN1056

CONTACTS AND LOCATIONS:
Locations (7):
- ARENSIA Exploratory Medicine LLC, Tbilisi, Georgia
- ARENSIA Exploratory Medicine Phase I Unit, Chisinau, Moldova
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - MD Anderson Cancer Centre, Madrid
  - Clinica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No